CLINICAL TRIAL: NCT05226455
Title: A Phase I-II Study to Assess Venetoclax + Azacitidine and Donor Lymphocyte Infusion in Patients With MDS or AML in Relapse After Allohematopoietic Stem Cell Transplantation
Brief Title: Venetoclax in Patients With MDS or AML in Relapse After AHSCT
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VENTOGRAFT; 2024-514877-23-00 (EU CTIS Number)
Record Dates: First submitted 2022-01-11; First posted 2022-02-07 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: MDS; AML
Keywords: MDS; AML; AHSCT; Venetoclax; Azacitidine; DLI
MeSH Terms: interventions — venetoclax; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- venetoclax + azacitidine +/- donor lymphocyte infusion (Experimental): Venetoclax + azacitidine +/- donor lymphocyte infusion (maximum 12 cycles). Venetoclax: on D1 to D14 of 28 days cycle ; Phase I: 4 dose levels: 50, 100, 200, 400 mg/d, starting dose at 100 mg ; Phase II: dose defined in the phase I.
  Azacitidine 75 mg/m²/d or 50 mg/m²/d (if allohematopoietic stem cell transplantation relapse < 4 months) x 5 days (on D1 to D5 of 28 days cycle).
  Interventions: Drug: venetoclax + azacitidine +/- donor lymphocyte infusion

INTERVENTIONS:
Drug: venetoclax + azacitidine +/- donor lymphocyte infusion — Venetoclax will be given once daily orally on days 1 to 14 for all cycles. Venetoclax + azacitidine +/- donor lymphocyte infusion (12 cycles maximum)
  Other Names: venclyxto; vidaza

SUMMARY:
Study to assess venetoclax + azacitidine and donor lymphocyte infusion (DLI) in patients with myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML) in relapse after allohematopoietic stem cell transplantation (AHSCT).

DETAILED DESCRIPTION:
A phase I-II study to assess venetoclax + azacitidine and donor lymphocyte infusion (DLI) in patients with myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML) in relapse after allohematopoietic stem cell transplantation (AHSCT).

ELIGIBILITY:
Inclusion Criteria:

1. Documented cytologic relapse of MDS according to FAB/WHO classification 2016 (including CMML with WBC < 13000/mm3) or AML, with WBC < 15000/mm3, after allo-SCT.

   Relapse of MDS or AML is defined as :
   * Return to pretreatment bone marrow blast percentage
   * Decrement of at least 50% from maximum remission
2. Age ≥ 18 years.
3. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
4. Patient must have adequate organ function:

   * Serum creatinine < 2 mg/dL or calculated creatinine clearance ≥ 30 mL/min for patients with creatinine levels > 1.5 times Upper Limit of Normal
   * Serum total bilirubin ≤ 2.5 times Upper Limit of Normal or direct bilirubin ≤ Upper Limit of Normal for patients with total bilirubin levels ≥ 2 mg/d
   * Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 2.5 times Upper Limit of Normal
   * Alkaline phosphatase ≤ 5 times Upper Limit of Normal (if > 2.5 times Upper Limit of Normal, then liver fraction should be ≤ 2.5 times Upper Limit of Normal).
5. Patient not refractory to platelet transfusions.
6. Female subject of childbearing potential must practice at least one protocol specified method of birth control, starting on Study Day 1 through at least 30 days after the last dose of venetoclax or 6 months after the last dose of azacitidine.

   Not being of childbearing potential is defined as:
   * Age > 55 years with no menses for 12 or more months without an alternative medical cause, or
   * Age ≤ 55 years with no menses for 12 or more months without an alternative medical cause AND an Follicle Stimulating Hormone (FSH) level > 40 IU/L, or
   * Permanent surgical sterility (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
7. Female subjects of childbearing potential must have negative results for pregnancy test performed:

   * At Screening with a serum sample obtained within 14 days prior to the first study drug administration, and
   * Prior to dosing with urine sample obtained on Cycle 1 Day 1, if it has been > 7 days since obtaining the serum pregnancy test results.

   Female subjects who are not of childbearing potential at Screening do not require pregnancy testing.
8. Male subjects sexually active with female partner(s) of childbearing potential, must agree from first dose of study drug(s) through at least 30 days after the last dose of venetoclax or 3 months after the last dose of azacitidine, whichever is later, to practice the protocol specified contraception.
9. Patient is available for periodic blood sampling, study related assessments, and appropriate clinical management at the treating institution for the duration of the study.
10. Patient has the ability to understand and willingness to sign an informed consent form indicating the investigational nature of the study.
11. Patient is able to swallow capsules.

Exclusion Criteria:

1. Patient has active and uncontrolled infection.
2. Patient has active acute or chronic Graft-versus-Host-Disease (GVHD).
3. Patient receives more than 1mg/kg/day prednisolone.
4. Patient has uncontrolled intercurrent illness or circumstances that could limit compliance with the study, including but not limited to the following: symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, pancreatitis, or psychiatric or social conditions that may interfere with patient compliance.
5. Patient is currently participating or has participated in a study with an investigational compound or device within 30 days of initial dosing with study drug.
6. Patient has known human immunodeficiency virus (HIV) infection or HIV-related malignancy.
7. Patient has clinically active hepatitis B or hepatitis C infection.
8. Patient has a known allergy or hypersensitivity to any component of venetoclax or azacitidine.
9. Patient with a "currently active" second malignancy, other than non-melanoma skin cancer and carcinoma in situ of the cervix, should not be enrolled. Patients are not considered to have a "currently active" malignancy if they have completed therapy for a prior malignancy, are disease free from prior malignancies for > 2 years or are considered by their physician to be at less than 30% risk of relapse.
10. Patient has received growth factors such as erythropoietin alfa (EPO) or granulocyte colony-stimulating factor (G-CSF) or has received non cytotoxic agents (including low dose oral chemotherapy) in the 30 days before inclusion. In case of previous cytotoxic treatment, an interval of 3 months is required.
11. Patient is on any systemic steroids that have not been stabilized to the equivalent of ≤ 10 mg/day prednisone during the 4 weeks prior to the start of the study drugs.
12. Patients with clinical evidence of Central Nervous System leukemia.
13. Patient has a history of Gastrointestinal surgery or other procedures that might interfere with the absorption or swallowing of the study drugs.
14. Subject has received strong or moderate CYP3A (Cytochrome P450, family 3, subfamily A) inhibitors within 3 days prior to the first dose of study drug.
15. Patient is unable to take and/or tolerate oral medications on a continuous basis.
16. Patient is pregnant or breastfeeding within the projected duration of the study.
17. Subject has a malabsorption syndrome or other condition that precludes an enteral route of administration.
18. Absence of social security.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2022-11-23 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Phase I: Dose-finding study | At the end of cycle 1 of venetoclax + azacitidine (each cycle is 28 days)
  Evaluation of Dose-limiting toxicity (DLT) to determine the optimal dose level in terms of both toxicity and safety for venetoclax + azacitidine
Phase II: Overall improvement rate of venetoclax + azacitidine +/- DLI | After 8 cycles of venetoclax + azacitidine (each cycle is 28 days)
  Response assessment performed according to modified IWG (International Working Group) 2006 criteria for myelodysplastic syndrome and to European Leukemia Net criteria for acute myeloid leukemia

SECONDARY OUTCOMES:
Toxicity assessment | At 60 months (at end of study)
  Adverse events analyzed by frequency, NCI CTCAE 5.0 grade, and causality
Graft-versus-Host-Disease (GVHD) rate | At 60 months (at end of study)
  Acute and chronic graft-versus-host-disease (GVHD) rate assessment (graft-versus-host events analyzed by frequency and grade)
Duration of response | At 60 months (at end of study)
  Duration of response defined as time from the date of the first observed response (complete or partial) to the date of first subsequent documented disease progression or relapse or death
Overall survival | At 60 months (at end of study)
  Overall Survival defined as time from the date of the first dose of venetoclax to the date of death or end of study
Progression-free survival | At 60 months (at end of study)
  Progression-free Survival for patients with at least a partial response defined as time from the date of the first dose of venetoclax to the date of the first documented disease progression or relapse or death
Event-free survival | At 60 months (at end of study)
  Event-free Survival defined as time from the date of the first dose of venetoclax to the date of earliest disease progression or death

OTHER OUTCOMES:
Correlation between patient overall mutational status before and after treatment | At 60 months (at end of study)
  Mutational analysis performed by NGS (next-generation sequencing) at screening and then at each protocol evaluation (post 4, 6 and 8 cycles of venetoclax + azacitidine and at end of study)
Prognostic impact of Minimal Residual Disease (MRD) on outcome | At 60 months (at end of study)
  Minimal Residual Disease (MRD) assessment by flow cytometry and allelic variant frequency (VAF) of baseline mutations

CONTACTS AND LOCATIONS:
Overall Officials: Thomas CLUZEAU, PHD, Principal Investigator — CHU de Nice - Hôpital l'Archet I
Locations (13):
- France (13):
  - CHU d'Amiens Picardie - Site sud, Amiens
  - CHU d'Angers, Angers
  - CHU de Grenoble, Grenoble
  - Hôpital Dupuytren, Limoges
  - Hôpital Saint-Eloi, Montpellier
  - CHU Hôtel Dieu, Nantes
  - Hôpital l'Archet I, Nice
  - Hôpital Saint louis, Paris
  - CHU de Haut-Lévèque, Pessac
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Centre Henri Becquerel, Rouen
  - Institut de Cancérologie de la Loire Lucien Neuwirth, Saint-Priest-en-Jarez
  - IUCT Oncopole, Toulouse